CLINICAL TRIAL: NCT04393714
Title: Demineralized Dentin Graft With Hydrochloric Acid Versus Nitric Acid in Alveolar Ridge Preservation. Randomised Controlled Clinical Trial
Brief Title: Demineralized Dentin Graft With Hydrochloric Acid Versus Nitric Acid in Alveolar Ridge Preservation
Acronym: DDG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed AbdelRaouf Hussein, Principal investigator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ARP2020
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Split-mouth prospective randomized clinical trial with 1:1 assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous dentin graft treated with nitric acid (Experimental)
  Interventions: Procedure: Alveolar ridge preservation after extraction
- autogenous dentin graft treated with hydrochloric acid (Active Comparator)
  Interventions: Procedure: Alveolar ridge preservation after extraction

INTERVENTIONS:
Procedure: Alveolar ridge preservation after extraction — atraumatic extraction followed by graft material insertion

SUMMARY:
The reduction in alveolar bone dimensions is an inevitable outcome after tooth extraction due to the healing events that results in bone modeling/remodeling. Alveolar ridge preservation is a successful approach that aids in reducing these changes greatly. Various techniques have been employed to achieve that outcome utilizing bone grafts and/or membrane. Dentin graft is a promising type that can overcome many of the limitations facing mainstream grafts. Autogenous source serve the advantage of providing graft with no cross-infection risk or immunogenicity. Moreover, the unique structure of dentin makes it suitable for osteoinduction and osteoconduction that yields favorite bone regeneration outcomes. Demineralization of dentin is essential to release trapped growth factors, expose collagen fibrils and enhance the grafts degradability and replacement by native tissues. Many acids have been investigated for the use in chairside preparation of the dentin graft and hence, clinicians are faced with different choices but little evidence regarding the acid which yield s better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable teeth
* medically healthy
* able to provide informed consent and attend follow-up period

Exclusion Criteria:

* pregnant
* smokers or alcoholic
* severe bone loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone changes | 6 months
  width and height losses (quantitative in mm)

SECONDARY OUTCOMES:
histological analysis | 6 months
  Histologic observations (qualitative) and histomorphometric measurements (quantitative in %)
soft tissue healing | Biweekly for 6 weeks
  rate of wound epitheliallization

IPD SHARING:
Plan to Share IPD: No